CLINICAL TRIAL: NCT01382446
Title: Evaluating Effectiveness of Chlorhexidine Gluconate Oral Care for Adults
Brief Title: Chlorhexidine Gluconate Oral Care for Adults Experiencing Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Madelon Petersen, Research Clinician, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#09NU127
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Trauma; Mechanical Ventilation; Ventilator Associated Pneumonia; Oral Care
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Wounds and Injuries | interventions — chlorhexidine gluconate; Toothpastes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Oral Care Regimen (Active Comparator): Current oral care protocol includes the use of 1.5% H2O2-coated swabs every four hours, toothbrushing with toothpaste every 12 hours, and use of continuous subglottic suction apparatus.
  Interventions: Other: Toothpaste
- Chlorhexidine Oral Care Regimen (Experimental): This study will compare our current oral care practice with the use of Chlorhexidine Gluconate 0.12% (Peridex, 3M Corporation) Twice daily in addition to regularly scheduled oral care as a means to decrease the incidence of VAP utilizing evidence-based strategies.
  Interventions: Drug: Chlorhexidine gluconate

INTERVENTIONS:
Drug: Chlorhexidine gluconate — 0.12% Chlorhexidine Gluconate 15ml Twice Daily, administered via toothbrushing and swabbing teeth, tongue, gingiva, and oral mucosa.
  Other Names: Peridex
  Arms: Chlorhexidine Oral Care Regimen
Other: Toothpaste — Brushing the teeth, tongue, gingiva, and oral mucosa twice daily with toothbrush and toothpaste.
  Arms: Standard Oral Care Regimen

SUMMARY:
Examine the use of 0.12% Chlorhexidine Gluconate as an adjunct to current oral care protocol for trauma patients on ventilator support to decrease the incidence of Ventilator Associated Pneumonia and oral bacterial load.

DETAILED DESCRIPTION:
To see a significant decrease in the bacterial load in the oral mucosa and subsequently, a decrease in the pathogenesis of Ventilator Associated Pneumonia through the use of an oral rinse containing 0.12% Chlorhexidine Gluconate as part of an oral care protocol. Current oral care protocol includes the use of 1.5% H2O2-coated swabs every four hours, toothbrushing with toothpaste every 12 hours, and use of continuous subglottic suction apparatus.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to ICUs located in Tower Two Critical Care Units: Medical, Surgical, Medical #2, and Trauma Intensive Care Units.
* Patients will be randomized to either treatment or standard group based on day of admission to Intensive Care Units. No limitation regarding gender, race, and ethnicity so that the sample will reflect "typical" Trauma population.

Exclusion Criteria:

* All patients admitted under "Doe" Status
* All patients with acute cervical spine injuries or facial fractures that oral care will create further harm to the patient (physician order stating "no oral care to be given" will be in chart)
* All patients with Oral Trauma or Oral Surgery
* All minors (Study will be completed in Adult Critical Care Units)
* Patients with allergy to chlorhexidine
* Patients without Teeth, or with fewer than 6 teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Thomas, MSN, Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited upon arrival to the Intensive Care Unit, or after mechanical ventilation was initiated.
Pre-assignment Details: Patients were randomized into groups after enrollment.
Groups:
- Standard Oral Care Regimen: Toothpaste : Brushing the teeth, tongue, gingiva, and oral mucosa twice daily with toothbrush and toothpaste.
- Chlorhexidine Oral Care Regimen: Chlorhexidine gluconate : 0.12% Chlorhexidine Gluconate 15ml Twice Daily, administered via toothbrushing and swabbing teeth, tongue, gingiva, and oral mucosa.
Period: Overall Study
Arm/Group | Standard Oral Care Regimen | Chlorhexidine Oral Care Regimen
Started | 33 | 33
Completed | 30 | 29
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Removal from Mechanical Ventilation | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Oral Care Regimen | Chlorhexidine Oral Care Regimen | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 25 | 57
  >=65 years | 1 | 8 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (16.279) | 45.5 (19.96) | 43.88 (18.355)
Gender [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 22 | 25 | 47
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Chlorhexidine Gluconate Oral Care for Trauma Patients
Description: Examination of number of participants who do not develop oral bacteria and Ventilator Associated Pneumonia when an oral rinse containing 0.12% Chlorhexidine Gluconate is used as part of a oral care protocol.
Time Frame: 18 Months
Population: Intention to Treat Analysis Used
Measure: Number; unit: participants
Arm/Group | Standard Oral Care Regimen | Chlorhexidine Oral Care Regimen
Number analyzed (Participants) | 33 | 33
participants | 30 | 29

ADVERSE EVENTS:
Arm/Group | Standard Oral Care Regimen | Chlorhexidine Oral Care Regimen
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

LIMITATIONS AND CAVEATS:
Enrolling of trauma patients - consenting patients with unknown identification or next of kin status led to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No